CLINICAL TRIAL: NCT06064110
Title: Pictou County PEP: A Phase 2 Trial of a Six-Month Home-Based Personal Empowerment Program to Improve the Mental and Physical Health of Adults With a Chronic Medical Condition Living in Pictou County
Brief Title: Pictou County PEP: A 6-Month, Home-Based, Personal Empowerment Program for Adults With a Chronic Medical Condition Living in Pictou County
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Dalhousie University (Other)
Responsible Party: Principal Investigator, Gabriela Ilie, Associate Professor, Dalhousie University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pictou-County-PEP
Record Dates: First submitted 2023-09-26; First posted 2023-10-03 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Chronic Condition
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental)
  Interventions: Behavioral: Pictou County Person Empowerment Program

INTERVENTIONS:
Behavioral: Pictou County Person Empowerment Program — The 6 month home-based program focuses on aerobic and strength training, meditation/relaxation techniques, social connection, and overall healthy lifestyle practices supported with daily email reminders. The aerobic (5 times/week) and strength (2 times/week) program will comprise of a single 30-minute session daily, the meditation/relaxation practice is 10 minutes daily, the intimacy and connection component consists of engaging in at least one form of intimacy practice prescribed, per day. Optional social connection components will be offered, such as pairing participants up with peers from the study, monthly Zoom videoconferences, and monthly in-person events in Pictou County to further promote healthy lifestyle habits.
  Other Names: PictouCountyPEP

SUMMARY:
The Pictou County Personal Empowerment Program is a comprehensive health promotion program aiming to improve the quality of life as well as both physical and mental health in Adults living with chronic medical conditions. The program includes daily email communications over 6 months that encourage a range of self-management and health promoting activities, including strength and aerobic exercise, yoga, stress reduction techniques, dietary improvements, relationship/intimacy education and more.

ELIGIBILITY:
INCLUSION CRITERIA:

* Age >18;
* Diagnosed with one or more chronic medical conditions, as per the participant's report, including but not restricted to the following (complete list in protocol appendix):

  * Heart disease / cardiovascular disease / stroke
  * High blood pressure
  * Diabetes including a diagnosis of pre-diabetes
  * Chronic respiratory disease
  * Chronic neurologic disease
  * Chronic kidney disease
  * Chronic liver disease
  * Immunodeficiency
  * Overweight or Obese (BMI >25)
  * Psychiatric or mental health issue - e.g., depression and anxiety
  * Substance-related and addictive disorders (e.g alcohol, smoking, etc.);
* Resident of Pictou County, Nova Scotia;
* Existing (or willingness to create) email account and willingness to access email daily;
* Ability to follow website links to watch YouTube videos;
* Ability to understand and speak English;
* Ability to participate in low to moderate levels of physical activity and strength training;
* Ability and willingness to fill out an online survey at baseline, and 6, 12 months, and fill in a weekly compliance survey for the six months of the program.

EXCLUSION CRITERIA:

* Diagnosed with cancer in the last 5 years and/or received treatment for cancer in the last 5 years;
* Myocardial infarction or stroke within the last year AND without written approval from their Family Physician, Cardiologist, or Study Physician that they are safe to exercise;
* Unable to access the internet daily during the intervention;
* Lack of access to a computer or smartphone to receive emails required for study intervention.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2023-11-24 (Actual); Primary Completion 2025-05-14 (Actual); Study Completion 2025-10-28 (Actual)

PRIMARY OUTCOMES:
Mental Health as assessed by the Kessler Kessler Psychological Distress Scale (K10) | 6-12 months
  A 10 item questionnaire that assesses psychological distress. The scale has a score range of 10-50, with higher scores indicating worse mental health.

SECONDARY OUTCOMES:
Incidence and severity of participant self-reported adverse events | 6-12 months
The Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) | 6-12 months
  A 40-item measure that assesses self-reported fatigue and its impact upon daily life, using a 5 point Likert-type scale with values ranging from 0-5, where higher scores represent worse outcomes.
Personality as assessed by the Ten-Item Personality Inventory (TIPI) | 6-12 months
  A 10 item questionnaire assessing the Big-Five personality dimensions (Extraversion, Agreeableness, Conscientiousness, Emotional Stability, Openness to Experiences). The scale has a score range of 1-14 for each dimension with higher scores indicating a higher level of that personality trait.
Alcohol Habit assessed by questions from the National Health Institute Alcohol Consumption questionnaire. | 6-12 months
  Questions assessing alcohol consumption using semantic differential scales that have a range of up to 11 response options. Response options range from never consuming alcohol to daily consumption, as well as consuming no alcohol each day to 25+ drinks a day on average, with higher scores being worse.
Smoking habit assessed by the Global Adult Tobacco Survey 2020 (GATS). | 6-12 months
  Questions assessing current and past smoking habit using semantic differential scales with possible answers ranging from daily smoking to not smoking at all. Lower scores indicate higher smoking habit/worse outcome.
Diet assessed by the Rapid Eating Assessment for Participants (REAP-S). | 6-12 months
  A 16 item questionnaire assessing diet quality. The scale has a score range of 13-39 with a higher score indicating a higher diet quality.
Comorbidity level assessed by the modified Charlson Comorbidity Index (CCI) | 6-12 months
  A 21 item questionnaire that uses a weighted index to assess the quantity and severity of comorbidities a patient has. Each comorbidity category has a related weight, ranging on a scale of 1-6, with higher scores representing worse outcomes.
Availability of social support assessed by the MOS Social Support Survey | 6-12 months
  A 19 item questionnaire that assesses emotional/informational support, positive social interaction, tangible support and affectionate support. Higher item scores reflect a higher level of social support.
Sleep Quality as assessed by the Pittsburgh Sleep Quality Index (PSQI) | 6-18 months
  A 19 item questionnaire that assesses sleep quality and disturbances. The scale has a score range of 0-21 with a higher score indicating worse sleep quality.
Sedentary behaviour measured by the Sedentary Behaviour Questionnaire (SBQ) for Adults. | 6-12 months
  Two 9 item questionnaires (weekday and weekend) with each item scored to none to 6 hours or more. The total score is the sum of the amount of time and as it increases it indicates higher amount of sedentary behaviour.
Anxiety severity assessed by the GAD-7. | 6-12 months
  A 7 item questionnaire with scores ranging from 0-21 higher scores indicating more severe level of anxiety.
Relationship satisfaction as assessed by the Dyadic Adjustment Scale (RDAS-14). | 6-12 months
  A 14 item questionnaire that measure an individual's perceptions of their relationship with an intimate partner. The scale has a total score range of 1-151 with a higher score indicating better satisfaction.
Center for Epidemiologic Studies Depression Scale (CES-D). | 6-12 months
  A 20 item questionnaire with a possible range of scores from zero to 60, with the higher scores indicating the presence of more depressive symptomatology.
Satisfaction with Life Scale (SWLS). | 6-12 months
  A 5 item questionnaire that was designed to measure subjective well-being. Scores range from 5-35 with higher scores indicating higher satisfaction with life.
Brief Illness Perception Questionnaire (BIPQ) | 6-12 months
  A 9 item scale that measures an individual's beliefs, feelings, and cognitive representations of one's illness. This questionnaire uses linear numeric scales with response options ranging from 0-10. Total scores can range from 0-80, with higher scores representing worse illness perceptions.
Perceived Stress Scale (PSS-10) | 6-12 months
  A 10-item scale that measures a person's perceived feelings of stress during the last month. This questionnaire uses a Likert-type scale with response options scores ranging from 0-4. Scores on the PSS-10 can range from 0-40 with higher scores indicating higher perceived stress.
WHO-5 Well-Being Index | 6-12 months
  A short, 5-item, generic global rating scale measuring subjective well-being using a Likert-type scale. Scores range from 0-5, with higher scores indicating better well-being.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Aberdeen Hospital, New Glasgow, Nova Scotia